CLINICAL TRIAL: NCT01439529
Title: Optimization of Response to Cardiac Resynchronization Therapy by Electrocardiogram: an Assessment of Medium-term Response
Brief Title: ECG Optimization of CRT: Evaluation of Mid-term Response
Acronym: BEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Elena Arbelo, Coordinator of the AF programme, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEST
Record Dates: First submitted 2011-09-19; First posted 2011-09-23 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: Cardiac; Resynchronization; Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nominal (Active Comparator): CRT device is programmed with the nominal values.
  Interventions: Other: Device programming: nominal
- Narrow QRS (Experimental): CRT device is programmed by QRS optimization
  Interventions: Other: Programming optimization by QRS

INTERVENTIONS:
Other: Device programming: nominal — CRT device is programmed to nominal values
  Arms: Nominal
Other: Programming optimization by QRS — CRT device is programmed by QRS optimization
  Arms: Narrow QRS

SUMMARY:
New simpler methods to optimize cardiac resynchronization therapy (CRT) are being evaluated, such as the use of the electrocardiogram.

In this prospective, double-blind, study, the investigators will evaluate:

Primary endpoint: To compare the clinical response to CRT in patients with the programming optimized by QRS versus the nominal suggested by the device.

Secondary endpoints:

1. To compare cardiac remodeling in patients with the programming optimized by QRS versus the nominal suggested by the device.
2. To evaluate the degree of asynchrony in both groups (nominal versus optimization by QRS) with respect to the intrinsic rhythm.
3. To evaluate the echocardiographic improvement in left ventricular (LV) filling in both groups.
4. To evaluate the differences in the optimal atrioventricular (AV) delay with atrial sensing or atrial pacing.

For that, 180 patients with an indication for CRT will be randomized to nominal programming of the device or optimization by the electrocardiogram for a narrower QRS. A clinical and echocardiographic evaluation will be done at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria: patients with standard indication of cardiac resynchronization

* Ejection fraction ≤35%.
* QRS duration ≥120 ms.
* New York Heart Association Functional Class 2-4..
* Left ventricular diameter ≥55 mm.
* Optimal medical treatment.

Exclusion Criteria:

* Patient refusal.
* Cardiopathy with a reversible cause.
* Prevision of heart transplantation.
* Atrial fibrillation.
* Complete AV block.
* AV delay >250 ms.
* Right bundle branch block.
* Severe peripheral vascular disease.
* Other diseases with < 1 year life expectancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-04; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Clinical response | 12 months
  Clinical response: survival without heart transplantation or death and >10% increased distance in the 6MWT.

SECONDARY OUTCOMES:
Echocardiographic response | 12 months
  Echocardiographic response: >15% decrease in LV end-systolic volume and survival without heart transplantation or death.
Pacing/sensing AV delay difference | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Arbelo, MD, PhD, Study Chair — Hospital Clinic Universitari de Barcelona; Lluís Mont, MD, PhD, Study Director — Hospital Clínic Universitari de Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Trucco E, Tolosana JM, Arbelo E, Doltra A, Castel MA, Benito E, Borras R, Guasch E, Vidorreta S, Vidal B, Montserrat S, Sitges M, Berruezo A, Brugada J, Mont L. Improvement of Reverse Remodeling Using Electrocardiogram Fusion-Optimized Intervals in Cardiac Resynchronization Therapy: A Randomized Study. JACC Clin Electrophysiol. 2018 Feb;4(2):181-189. doi: 10.1016/j.jacep.2017.11.020. Epub 2018 Feb 1. PMID 29749935